CLINICAL TRIAL: NCT03721289
Title: Evaluation in Real World of Molecular Testing and Treatment Patterns for EGFR Mutations in Patients With Advanced or Metastatic NSCLC at Front-line and Progression
Brief Title: Evaluation in Real World of Molecular Testing and Treatment Patterns for EGFR Mutation in Lung Cancer Patients
Acronym: PANORAMRETRO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00143
Record Dates: First submitted 2018-10-02; First posted 2018-10-26 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: All registered cases of stage IV NSCLC patients, treatment naïve, diagnosed in the participant institution during one year (from Jan 1st 2017 to Dec 31st 2017).
- Cohort 2: All EGFR positive patients progressed to an EFGR-TKI in the same period of time (from Jan 1st 2017 to Dec 31st 2017)

SUMMARY:
Evaluate molecular testing and treatment patterns for EGFR mutation in two different cohorts of stage IV NSCLC, at diagnosis (treatment naïve) and at the moment of progression to EGFR-TKIs. This study is non-indication seeking (NIS), descriptive in nature and does not attempt to test any specific a priori hypotheses.

DETAILED DESCRIPTION:
Objectives and Hypotheses : The objectives of this study are to evaluate molecular testing and treatment patterns for EGFR mutation in two different cohorts of stage IV NSCLC, at diagnosis (treatment naïve) and at the moment of progression to EGFR-TKIs. This study is non-indication seeking (NIS), descriptive in nature and does not attempt to test any specific a priori hypotheses. The following study objectives will be assessed:

Primary Objectives

* To estimate parameters associated with molecular testing patterns at diagnosis of advance disease and progression to EGFR TKIs
* To estimate parameters associated with treatment patterns at frontline and at progression to a EGFR TKI therpay

Secondary Objectives

* To estimate the rate of central nervous system (CNS) metastases at diagnosis and after disease progression in EGFR+ NSCLC patients
* To estimate parameters associated with biopsy related complications

Study Design This will be an observational retrospective study of patients with Stage IV NSCLC in two different cohorts from participating sites in Uruguay, Argentina, Costa Rica, Colombia, Chile, Peru, and Republica Dominicana. Cohort 1: newly diagnosed Stage IV NSCL who are treatment naive Cohort 2: stage IV NSCLC EGFRm progressed after first or second generation EGFR-TKI

Data of patients meeting the study inclusion/exclusion criteria will be collected from diagnosis of Satge IV (cohort 1) or diagnosis of progression after first or second generation EGFR-TKI (cohort 2) until the maximum follow up registered in the medical record.

Data will be collected and entered in the electronic case report form (eCRF). All data will be collected using patient medical records. The investigator will be responsible for ensuring that all the required data is collected and entered into the eCRF. The site will collect the data that will be uploaded according to the data entry procedures.

Study Population Cohort

1: all registered cases of stage IV NSCLC patients, treatment naïve, diagnosed in the participant institution during one year (from Jan 1st 2017 to Dec 31st 2017). Cohort 2: all EGFR positive patients progressed to an EFGR-TKI in the same period of time (from Jan 1st 2017 to Dec 31st 2017)

In the case one patient meets eligibility criteria for both cohorts, this patient will be included only in the EFGR-TKI progressed cohort.

Exposures There are no specific drug exposures or interventions being evaluated, as cohort eligibility is not exposure-based, but rather disease-based.

Study Measures

* Patient demographic and clinical characteristics
* Molecular testing rates at Stage IV and at progression to EGFR TKI
* Molecular testing EGFR mutation results (common/uncommon mutations at advanced diagnosis, and T790M at progression)
* Treatment patterns at frontline and progression to EGFR TKIs
* Biopsy-related complications
* Percentage of patinets presenting with CNS metastasis at diagnosis of stage IV and at progression to EGFR TKIsCNS

Sample:

All patients diagnosed with Stage IV NSCLC at diagnosis and at progression to an EGFR-TKI; from January 1st , 2017 to December 31st, 2017 in selected centers of Uruguay, Argentina, Chile, Colombia

Statistical Analysis No formal hypothesis testing is specified. Study measures including patient demographics and clinical characteristics, molecular testing rates and patterns, treatment patterns. Continuous study measures (e.g., age) will be reported descriptively with mean, standard deviation, median, minimum and maximum. Frequencies and percentages will be used to document categorical measures of interest (e.g., number and proportion of patients with a molecular test, number and proportion of patients with a EGFR mutation) and will include 95% CIs for key outcome variables.

Study Duration Estimated date of First Patient Data In: Q3 2018

Estimated date of Data Base Lock: Q1 2019

ELIGIBILITY:
Inclusion Criteria Cohort 1

* Adult male or female patients ≥ 18 years of age
* Newly diagnosed patients with stage IV NSCLC who are treatment naïve, from 1st Jan 2017 to Dec 31st 2017
* For patients still avile, provision of written informed consent as per local regulations

Cohort 2

* Adult male or female patients ≥ 18 years of age
* Patinets Stage IV NSCLC progressed after a first line TKI from 1st Jan 2017 to Dec 31st 2017.
* For patients still avile, provision of written informed consent as per local regulations

In the case one patient meets eligibility criteria for both cohorts, this patient will be included only in the EFGR-TKI progressed cohort.

Exclusion Criteria

• There are not exclusion criteria to this study. For an overview on the guidelines to determine disease progression, refer to Appendix A (Section 11).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: all registered cases of stage IV NSCLC patients, treatment naïve, diagnosed in the participant institution during one year (from Jan 1st 2017 to Dec 31st 2017).
  Cohort 2: all EGFR positive patients progressed to an EFGR-TKI in the same period of time (from Jan 1st 2017 to Dec 31st 2017) In the case one patient meets eligibility criteria for both cohorts, this patient will be included only in the EFGR-TKI progressed cohort.
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the EGFR mutation | Clinical charts from January 2013-december 2017
  Test used to determine EGFRm, registered in clinical charts

CONTACTS AND LOCATIONS:
Overall Officials: Florencia Reinhold, MD, Principal Investigator — AstraZeneca
Locations (10):
- Argentina (4):
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
- Research Site, Santiago, Chile
- Colombia (4):
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Medellín
  - Research Site, Montería
- Research Site, Montevideo, Uruguay